CLINICAL TRIAL: NCT02077725
Title: Measure the Impact of an Interdisciplinary Polypharmacy Clinic Within a Patient-entered Medical Home
Brief Title: Measuring the Impact of an Interdisciplinary Polypharmacy Clinic Within a Patient-centered Medical Home
Status: Withdrawn | Type: Observational
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Stuart Beatty, Assistant Professor of Clinical Pharmacy, Ohio State University
Other Study IDs: 2012H0067
Record Dates: First submitted 2014-03-02; First posted 2014-03-04 (Estimated); Last update posted 2022-09-30 (Actual); Status verified 2022-09

CONDITIONS: Polypharmacy
Keywords: drug related problems; comprehensive medication review; quality of life

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Interdisciplinary polypharmacy clinic: Patients will be seen in the interdisciplinary polypharmacy clinic for a complete comprehensive medication review
  Interventions: Other: interdisciplinary polypharmacy clinic visit

INTERVENTIONS:
Other: interdisciplinary polypharmacy clinic visit

SUMMARY:
Title: Measuring the impact of an interdisciplinary polypharmacy clinic within a patient-centered medical home

Objectives:

The primary objective of this project will be to track the types of interventions made in an interdisciplinary polypharmacy clinic to improve medication regimens and medication burden. Polypharmacy has been well documented in the literature as a risk for medication errors, adverse drug events, and morbidity. Team visits, including complete medication reviews, by pharmacists and physicians within a National Committee for Quality Assurance (NCQA) tier 3 patient-centered medical home (PCMH) at an academic medical center, can improve medication regimens. Secondary objectives include (1) measuring each patient's quality of life at baseline and one month post-intervention and (2) tracking the cost of medication additions and discontinuations.

Methods:

Patients taking ten or more chronic medications will be identified for referral to the polypharmacy clinic from a report generated from the electronic medical record. The polypharmacy clinic will be staffed by a pharmacist and medical resident with oversight from an attending physician who specializes in geriatrics. Drug-related problems identified during the visit will be resolved and categorized based upon indication, efficacy, cost, safety, and compliance. The numbers and types of interventions made, both during the primary visit and anticipated in the future, will be tracked. The 12-item short form (SF-12) survey will also be administered at baseline and one month post intervention. The increase or decrease in cost for medications added and removed during these visits will be captured using the average wholesale prices.

Preliminary Results Using descriptive statistics, the types of drug-related problems identified and interventions made will be reported. Changes in quality of life and monthly medication costs will also be described.

ELIGIBILITY:
Inclusion Criteria:

* Patients on 10 or more chronic medications
* Age 18 or older

Exclusion Criteria:

* Non-English speaking patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients within the general internal medicine patient-centered medical homes of The Ohio State University Division of General Internal Medicine
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2013-12; Primary Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Number and types of drug related problems identified | 1 year

SECONDARY OUTCOMES:
Assess quality of life at baseline and one month post polypharmacy clinic visit | 1 month
Cost of medication additions and discontinuations | 1 month

CONTACTS AND LOCATIONS:
Locations (1):
- The Ohio State University Division of General Internal Medicine Martha Morehouse, Columbus, Ohio, United States